CLINICAL TRIAL: NCT06886061
Title: Effect of Continuous Intake of Ergothioneine-containing Supplements on Skin Condition: a Randomized, Double Blind, Placebo-controlled Study
Brief Title: Effect of Continuous Intake of Ergothioneine-containing Supplements on Skin Condition
Acronym: EGTCLINIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai EGT Synbio Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UMIN000055792
Record Dates: First submitted 2025-03-03; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Skin
Keywords: Ergothioneine; Skin; Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Group (Placebo Comparator): The placebo group continuously ingests capsules without Ergothioneine over a period of 8 weeks.
  Interventions: Dietary Supplement: The capsules do not contain Ergothioneine.
- Ergothioneine Group (Experimental): The Ergothioneine group continuously ingests one capsule containing 30mg of Ergothioneine per day over a period of 8 weeks.
  Interventions: Dietary Supplement: The capsules contain Ergothioneine.

INTERVENTIONS:
Dietary Supplement: The capsules contain Ergothioneine. — Take one 30 mg Ergothioneine capsule orally every day for a period of eight weeks.
  Arms: Ergothioneine Group
Dietary Supplement: The capsules do not contain Ergothioneine. — Take one capsule devoid of Ergothioneine orally every day for a period of eight weeks.
  Arms: Placebo Group

SUMMARY:
This trial employed a non-randomized, double-blind, placebo-controlled design to evaluate the effects of DR. ERGO® Capsules (each containing 30mg of ergothioneine) on the skin condition of women aged 35 to 59 after continuous daily intake for 8 weeks. The trial assessed skin condition across multiple dimensions, including brightness, color tone, melanin, erythema, gloss, elasticity, and spots, using various instruments and questionnaire surveys. Additionally, safety was monitored through daily log records and safety evaluations.

DETAILED DESCRIPTION:
Ergothioneine (EGT), a naturally occurring amino acid-like antioxidant, was first discovered in Clavieps purpurea in 1909. It is widely found in mushrooms, legumes, and certain animal tissues. Studies have shown that ergothioneine protects skin cells by scavenging free radicals and reducing oxidative stress, thereby delaying skin aging. Additionally, it can inhibit melanin production, improve uneven skin tone, enhance the skin barrier function, and boost skin elasticity and radiance. In recent years, with growing attention to nutricosmetics, ergothioneine has gained significant interest for its potential anti-aging and skin-enhancing benefits.

The trial employed a non-randomized, double-blind, placebo-controlled design, adhering to the principles of the Helsinki Declaration and relevant Japanese ethical guidelines, and received approval from an ethics review committee. The primary objective of the study was to evaluate the effects of daily consumption of one DR. ERGO® capsule (each containing 30mg of ergothioneine) on the skin condition of women aged 35 to 59 over an 8-week period.

The trial design included strict inclusion and exclusion criteria to ensure consistency in the health status and testing conditions of the participants. During the trial, participants were required to maintain their normal lifestyle habits and avoid using any medications or cosmetics that might affect their skin condition. The study assessed skin condition across multiple dimensions-including brightness, color tone, melanin levels, erythema, gloss, elasticity, spots, and wrinkles-using various instruments and questionnaires. Additionally, safety was monitored through diary logs and safety assessments.

ELIGIBILITY:
Inclusion Criteria:

① Healthy women aged 35 to 59 years old.

② Individuals who feel that their skin condition is deteriorating (loss of radiance, dullness, pigmentation spots, etc.).

Exclusion Criteria:

* Individuals with a history of food allergies.

  * Pregnant or breastfeeding individuals.

    * Individuals with inflammation or wounds on their face.

      * Individuals taking medication that could affect the trial. ⑤ Individuals consuming health supplements that could affect the trial.

        ⑥ Individuals currently undergoing medical treatment or receiving prescriptions from a doctor.

        ⑦ Individuals undergoing hormone therapy.

        ⑧ Individuals with eyelash extensions, permanent eyeliner, or other forms of cosmetic tattooing around the eyes.

        ⑨ Individuals who have participated in human clinical trials within the last month or plan to do so during the trial period.

        ⑩ Individuals deemed unsuitable by the principal investigator of the trial.

Ages: 35 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2024-10-09 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Brightness & Color | Before the trial begins, at 4 weeks, and at 8 weeks.
  Using the SPECTRO PHOTOMETER NF555 (Japan Electric Color Industry Co., Ltd.), measure the brightness and color at the intersection points of vertical lines below both outer canthi and horizontal lines from the alae nasi. The L*a*b* method is used to measure L* value (brightness), a* value, and b* value (color). Higher values indicate brighter or more intense colors.
Melanin | Before the trial begins, at 4 weeks, and at 8 weeks.
  Using the Mexameter® MX 18 (Courage+Khazaka electronic GmbH), measure melanin at the same facial points as above to assess the content of melanin.
Erythema | Before the trial begins, at 4 weeks, and at 8 weeks.
  Using the Mexameter® MX 18 (Courage+Khazaka electronic GmbH), measure erythema at the same facial points as above to assess the content of erythema.
Gloss (Shine) | Before the trial begins, at 4 weeks, and at 8 weeks.
  Using the Glossymeter GL200MP (Courage+Khazaka electronic GmbH), measure the gloss at the specified facial points. This device measures true gloss unaffected by skin surface texture or color.
Elasticity | Before the trial begins, at 4 weeks, and at 8 weeks.
  Using the Cutometer® MPA580 (Courage+Khazaka electronic GmbH), measure elasticity at the designated facial points. Skin elasticity is evaluated through R2 (total elasticity), R5 (net elasticity), and R7 (elasticity upon retraction) ratios.
Spots | Before the trial begins, at 4 weeks, and at 8 weeks.
  Using VISIA® Evolution (Canfield Scientific Inc.), measure spots on both sides of the face at the defined locations. Assess the number of spots.

SECONDARY OUTCOMES:
Skin Condition | Before the trial begins, at 4 weeks, and at 8 weeks.
  Conduct three surveys before the trial begins, and at 4 and 8 weeks into the trial, covering 11 items: "moisture," "dryness," "softness," "gloss," "smoothness," "skin allergy condition," "texture," "makeup adherence," "tightness," "wrinkles," "transparency," "tightness after washing," "brightness," and overall skin satisfaction. Participants rate these aspects on a 9-point scale ranging from "very poor" to "very good."

CONTACTS AND LOCATIONS:
Overall Officials: Kaneko Takeshi, Principal Investigator — Japan Clinical Trial Association
Locations (1):
- Japan Clinical Trial Association N.A., Tokyo, Shinjukuku, Japan